CLINICAL TRIAL: NCT01013649
Title: A Phase II-R and a Phase III Trial Evaluating Both Erlotinib (Ph II-R) and Chemoradiation (Ph III) as Adjuvant Treatment for Patients With Resected Head of Pancreas Adenocarcinoma
Brief Title: Gemcitabine Hydrochloride With or Without Erlotinib Hydrochloride Followed by the Same Chemotherapy Regimen With or Without Radiation Therapy and Capecitabine or Fluorouracil in Treating Patients With Pancreatic Cancer That Has Been Removed by Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01987; NCI-2011-01987 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11-00773; CDR0000659092; RTOG 0848; RTOG-0848 (Other: NRG Oncology); RTOG-0848 (Other: CTEP); U10CA021661 (NIH); U10CA180830 (NIH); U10CA180868 (NIH)
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Results first posted 2024-10-24 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Adenocarcinoma; Pancreatic Ductal Adenocarcinoma; Pancreatic Intraductal Papillary-Mucinous Neoplasm; Stage I Pancreatic Cancer AJCC v6 and v7; Stage II Pancreatic Cancer AJCC v6 and v7
MeSH Terms: conditions — Pancreatic Intraductal Neoplasms | interventions — Radiotherapy, Conformal; Specimen Handling; Capecitabine; Drug Therapy; Erlotinib Hydrochloride; Fluorouracil; dehydroftorafur; Gemcitabine; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm I (gemcitabine hydrochloride or combination chemotherapy) (Active Comparator): Patients receive either gemcitabine hydrochloride or allowable combination chemotherapy per standard of care for 5 months. Patients undergo CT, MRI, and/or x-ray imaging throughout the trial. Patients also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline.
  Interventions: Procedure: Biospecimen Collection; Drug: Chemotherapy; Procedure: Computed Tomography; Drug: Gemcitabine Hydrochloride; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Procedure: X-Ray Imaging
- Arm II (gemcitabine hydrochloride, erlotinib hydrochloride) (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes once a week for 3 weeks then off 1 week and erlotinib hydrochloride PO once daily on days 1-28. Treatment repeats every 28 days for up to 5 courses in the absence of disease progression or unacceptable toxicity. Patients undergo CT, MRI, and/or x-ray imaging throughout the trial. Patients also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline. (closed to accrual 4/2/14)
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Erlotinib Hydrochloride; Drug: Gemcitabine Hydrochloride; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Procedure: X-Ray Imaging
- Arm III (chemotherapy) (Experimental): Patients receive the same treatment as in arm I for 1 month. Patients undergo CT, MRI, and/or x-ray imaging throughout the trial. Patients also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline.
  Interventions: Procedure: Biospecimen Collection; Drug: Chemotherapy; Procedure: Computed Tomography; Drug: Gemcitabine Hydrochloride; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Procedure: X-Ray Imaging
- Arm IV (chemotherapy, chemoradiotherapy) (Experimental): Patients receive the same treatment as in arm I for 1 month. Beginning within 7-21 days after completion of chemotherapy, patients undergo radiotherapy (3-dimensional conformal radiotherapy or intensity-modulated radiotherapy) 5 days per week for 5.5 weeks (28 fractions). During radiotherapy, patients receive either capecitabine PO BID 5 days per week or fluorouracil IV continuously for 5.5 weeks or until radiotherapy is completed. Patients undergo CT, MRI, and/or x-ray imaging throughout the trial. Patients also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Biospecimen Collection; Drug: Capecitabine; Drug: Chemotherapy; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Gemcitabine Hydrochloride; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Procedure: X-Ray Imaging

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3-dimensional conformal radiation therapy
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D radiotherapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal; Three dimensional external beam radiation therapy (procedure)
  Arms: Arm IV (chemotherapy, chemoradiotherapy)
Procedure: Biospecimen Collection — Undergo blood and tissue sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
  Arms: Arm IV (chemotherapy, chemoradiotherapy)
Drug: Chemotherapy — Given combination chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
  Arms: Arm I (gemcitabine hydrochloride or combination chemotherapy); Arm III (chemotherapy); Arm IV (chemotherapy, chemoradiotherapy)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: CP 358; CP-358; Cp-358,774; CP358; OSI 774; OSI-774; OSI774; Tarceva
  Arms: Arm II (gemcitabine hydrochloride, erlotinib hydrochloride)
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: Arm IV (chemotherapy, chemoradiotherapy)
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011
Radiation: Intensity-Modulated Radiation Therapy — Undergo intensity-modulated radiation therapy
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
  Arms: Arm IV (chemotherapy, chemoradiotherapy)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: X-Ray Imaging — Undergo x-ray imaging
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This randomized phase II-R/III trial studies gemcitabine hydrochloride with or without erlotinib hydrochloride followed by the same chemotherapy regimen with or without radiation therapy and capecitabine or fluorouracil in treating patients with pancreatic cancer that was removed by surgery. Drugs used in chemotherapy, such as gemcitabine hydrochloride, capecitabine, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays to kill tumor cells. Giving chemotherapy together with or without erlotinib hydrochloride and/or radiation therapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether chemotherapy is more effective when given with or without erlotinib hydrochloride and/or radiation therapy in treating pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the addition of erlotinib (erlotinib hydrochloride) to gemcitabine (gemcitabine hydrochloride) adjuvant chemotherapy shows a signal for improved survival as compared to gemcitabine alone following R0 or R1 resection of head of pancreas adenocarcinoma (including adenocarcinoma of the head, neck, and uncinate process). (Phase II-R) II. To determine whether the use of concurrent fluoropyrimidine and radiotherapy following adjuvant gemcitabine based chemotherapy or non-gemcitabine based chemotherapy such as modified fluorouracil-leucovorin-irinotecan-oxaliplatin regimen (FOLFIRINOX) further enhances survival for such patients who are without evidence of progressive disease after 5 months of adjuvant chemotherapy. (Phase III)

SECONDARY OBJECTIVES:

I. To evaluate disease-free survival of adjuvant chemotherapy followed by radiotherapy and concurrent fluoropyrimidine for patients with resected head of pancreas adenocarcinoma who are disease free after 5 months of adjuvant chemotherapy.

II. To evaluate disease-free survival of standard adjuvant gemcitabine chemotherapy with and without erlotinib for patients with resected head of pancreas adenocarcinoma.

III. To evaluate adverse events with and without erlotinib for patients with resected head of pancreas adenocarcinoma.

IV. To evaluate adverse events of adjuvant chemotherapy with or without radiation therapy and concurrent fluoropyrimidine for patients with resected head of pancreas adenocarcinoma who are disease free after adjuvant chemotherapy.

V. To evaluate preoperative cross-sectional imaging of the primary head of pancreas adenocarcinoma in order to determine the frequency with which objective criteria of resectability are present.

VI. To determine if patients reporting low baseline fatigue, as measured by the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue, predicts survival and to explore correlations between baseline fatigue, as measured by Patient-Reported Outcomes Measurement Information System (PROMIS), and survival.

OUTLINE: Patients without disease progression after treatment in arm I or II are randomized to 1 of 2 additional treatment arms (arm III or IV).

ARM I: Patients receive either gemcitabine hydrochloride or allowable combination chemotherapy per standard of care for 5 months.

ARM II (closed to accrual 4/2/14): Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes once a week for 3 weeks then off 1 week and erlotinib hydrochloride orally (PO) once daily on days 1-28. Treatment repeats every 28 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.

ARM III: Patients receive the same treatment as in arm I for 1 month.

ARM IV: Patients receive the same treatment as in arm I for 1 month. Beginning within 7-21 days after completion of chemotherapy, patients undergo radiotherapy (3-dimensional conformal radiotherapy or intensity-modulated radiotherapy) 5 days per week for 5.5 weeks (28 fractions). During radiotherapy, patients receive either capecitabine PO twice daily (BID) 5 days per week or fluorouracil IV continuously for 5.5 weeks or until radiotherapy is completed.

Patients undergo computed tomography (CT), magnetic resonance imaging (MRI), and/or x-ray imaging throughout the trial. Patients also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline.

After completion of study treatment, patients are followed up every 3-6 months for up to 4 years, then yearly.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of primary head of pancreas invasive adenocarcinoma managed with a potentially curative resection (i.e., removal of all gross tumor) involving a classic pancreaticoduodenectomy (Whipple) or a pylorus preserving pancreaticoduodenectomy; patients with invasive adenocarcinoma that also contains a component of intraductal papillary mucinous neoplasm (IPMN) are eligible

  * The operating surgeon must document in the operative note that a complete gross excision of the primary tumor was achieved; the pathology report must include documentation of the margin status and the size of the tumor; the pathology report must also include the status of the three major margins-bile duct, pancreatic parenchyma, and retroperitoneal (uncinate)
* For patients who have not started their chemotherapy prior to registration, the interval between definitive tumor-related surgery and 1st step registration must be between 21-70 days; for patients entering on the study who have already received up to 3 months of adjuvant chemotherapy as per the treating institution, the interval between definitive tumor-related surgery and day one of adjuvant chemotherapy must be between 21-77 days
* Patients will be staged according to the 6th edition American Joint Committee on Cancer (AJCC) staging system with pathologic stage T1-3, N0-1, M-0 being eligible. Pathologic reporting using the College of American Pathologists (CAPS) format is strongly encouraged
* Age >= 18
* Zubrod performance status 0 or 1
* Complete history and physical examination including weight and Zubrod status within 31 days of study entry (or within 31 days prior to day 1 of chemotherapy post-surgery for those patients having started chemotherapy prior to first step registration)
* Before starting therapy the patient should be able to maintain adequate oral nutrition of >= 1500 calories estimated caloric intake per day and be free of significant nausea and vomiting
* Complete blood count (CBC)/differential obtained within 21 days of registration on study (or within 21 days prior to day 1 of chemotherapy post-surgery for those patients having started chemotherapy prior to first step registration)
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 8.0 g/dL (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 8.0 g/dl is acceptable)
* Post resection serum cancer antigen (CA)19-9 =< 180 units/mL AND prior to any systemic treatment
* Serum total bilirubin =< twice the institutional upper limit of normal (ULN) within 21 days of registration on study (or within 21 days prior to day 1 of chemotherapy post-surgery for those patients having started chemotherapy prior to first step registration)
* Creatinine levels =< twice the institutional upper limit of normal within 21 days of registration on study (or within 21 days prior to day 1 of chemotherapy post-surgery for those patients having started chemotherapy prior to first step registration)
* Serum glutamic oxaloacetic transaminase (SGOT) must be =< 2.5 x the institutional upper limit of normal within 21 days of registration on study (or within 21 days prior to day 1 of chemotherapy post-surgery for those patients having started chemotherapy prior to first step registration)
* Negative serum pregnancy test for women of childbearing potential within 14 days of study registration
* Abdominal/pelvic CT scan with contrast is preferred; abdominal CT alone is acceptable only if insurance restrictions are experienced; chest CT/x-ray (CT of chest preferred) within 31 days of registration on study (or within 31 days prior to day 1 of chemo post-surgery for those patients having started chemotherapy prior to first step registration); patients allergic to IV contrast can have MRI of the abdomen/pelvis instead
* Signed study-specific informed consent
* Consultation, agreement, and documentation in the patient's chart by a radiation oncologist that patient is suitable to receive radiotherapy per this protocol
* Women of childbearing potential and male participants must practice adequate contraception
* Patients with active human immunodeficiency virus (HIV) infection are eligible if their cluster of differentiation (CD)4 count is > 499/cu mm and their viral load is < 50 copies/ml; use of highly active antiretroviral treatment (HAART) is allowed

Exclusion Criteria:

* Patients with non-adenocarcinomas, adenosquamous carcinomas, islet cell (neuroendocrine) tumors, cystadenomas, cystadenocarcinomas, carcinoid tumors, duodenal carcinomas, distal bile duct, and ampullary carcinomas; patients with tumors that are largely intraductal papillary mucinous neoplasms (IPMN) with a minimal or minor component of invasive carcinoma are not eligible; patients with acinar carcinomas are not eligible; patients with IPMN's that contain some secondary (minor) foci of adenocarcinoma are also not eligible
* Patients managed with a total pancreatectomy, a distal pancreatectomy, or central pancreatectomy
* Patients entering on the study after pancreaticoduodenectomy, who have not already started chemotherapy must not have had prior systemic chemotherapy for pancreas cancer; note that prior chemotherapy for a different cancer is allowable; for patients entering on the study who have already received up to 3 months of adjuvant chemotherapy as per the treating institution, patients must not have received adjuvant chemotherapy with agents other than gemcitabine, nab-paclitaxel, oxaliplatin, fluoropyrimidine, or irinotecan for the current pancreatic cancer; prior chemotherapy for a different cancer is allowable
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Previous history of invasive malignancy (except non-melanoma skin cancer) unless the patient has been disease free for at least 2 years prior to study entry (or first day of chemotherapy for patients having started chemotherapy prior to first step registration); patients with a previous history of carcinoma in situ are eligible
* Severe, active co-morbidity, defined as follows per time points indicated below (or per time points indicated below prior to the first day of chemotherapy for patients having started chemotherapy prior to first step registration):

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the 3 months of study registration
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
* Pregnant or lactating women
* Women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic
* If surgical margin status cannot be determined after consultation with the operating surgeon and the institutional pathologist, the patient will be ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2010-04-05 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2025-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross A Abrams, Principal Investigator — NRG Oncology
Locations (689):
- United States (678):
  - Providence Hospital, Mobile, Alabama
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Community Cancer Institute, Clovis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Saint Agnes Medical Center, Fresno, California
  - Marin General Hospital, Greenbrae, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - El Camino Hospital, Mountain View, California
  - Wilma Chan Highland Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Mercy General Hospital Radiation Oncology Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Hartford HealthCare - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - William Backus Hospital, Norwich, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Jackson Memorial Hospital-Holtz Children's Hospital, Miami, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Florida Cancer Affiliates, Trinity, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Saint John's Hospital, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Saint Anne's Hospital, Fall River, Massachusetts
  - Berkshire Medical Center - Cancer Center, Pittsfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Huron Valley-Sinai Hospital, Commerce, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Elliot Hospital, Manchester, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - New York Oncology Hematology PC - Albany, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Sands Cancer Center, Canandaigua, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Garnet Health Medical Center, Middletown, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Wilmot Cancer Institute Radiation Oncology at Greece, Rochester, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - East Carolina University, Greenville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Radiation Oncology Center, Alliance, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Salem Regional Medical Center, Salem, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Mid-Columbia Medical Center/Celilo Cancer Center, The Dalles, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Crozer-Chester Medical Center, Upland, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Radiation Oncology Associates Incorporated, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Carolina Blood and Cancer Care Associates PA, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Texas Oncology-Arlington South, Arlington, Texas
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Texas Oncology Bedford, Bedford, Texas
  - Texas Oncology - Denison Cancer Center, Denison, Texas
  - Texas Oncology-Flower Mound, Flower Mound, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Texas Oncology - Lewisville, Lewisville, Texas
  - Texas Oncology-Longview Cancer Center, Longview, Texas
  - Texas Oncology-McKinney, McKinney, Texas
  - Texas Oncology-Seton Williamson, Round Rock, Texas
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - Cancer Care Centers of South Texas- Northeast, San Antonio, Texas
  - Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Deke Slayton Cancer Center, Webster, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Belgium (4):
  - Hospital Univ. Erasme, Brussels
  - University Hospital Saint Luc, Brussels
  - Algemeen Ziekenhuis Groeninge Campus Kennedylaan, Kortrijk
  - AZ Turnhout-Campus Saint Elizabeth, Turnhout
- Canada (4):
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Ottawa Hospital-Civic Campus, Ottawa, Ontario
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
- Israel (3):
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky

REFERENCES:
- [Derived] Jethwa KR, Kim E, Berlin J, Anker CJ, Tchelebi L, Abood G, Hallemeier CL, Jabbour S, Kennedy T, Kumar R, Lee P, Sharma N, Small W Jr, Williams V, Russo S. Executive Summary of the American Radium Society Appropriate Use Criteria for Neoadjuvant Therapy for Nonmetastatic Pancreatic Adenocarcinoma: Systematic Review and Guidelines. Am J Clin Oncol. 2024 Apr 1;47(4):185-199. doi: 10.1097/COC.0000000000001076. Epub 2023 Dec 22. PMID 38131628
- [Derived] Conroy T, Lambert A, Ducreux M. Adjuvant and neoadjuvant approaches in pancreatic cancer. Curr Opin Oncol. 2023 Jul 1;35(4):326-333. doi: 10.1097/CCO.0000000000000962. Epub 2023 May 12. PMID 37222189
- [Derived] Batukbhai B, Herman JM, Zahurak M, Laheru DA, Le DT, Wolfgang CL, Zheng L, De Jesus-Acosta A. Survival Outcomes of Adjuvant Chemotherapy Combined With Radiation Versus Chemotherapy Alone After Pancreatectomy for Distal Pancreatic Adenocarcinoma: A Single-Institution Experience. Pancreas. 2021 Jan 1;50(1):64-70. doi: 10.1097/MPA.0000000000001724. PMID 33370024

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Gemcitabine Hydrochloride or Combination Chemotherapy): Patients receive either gemcitabine hydrochloride or [starting 06-28-2016] allowable combination chemotherapy per standard of care for 5 months. Patients undergo CT, MRI, and/or x-ray imaging throughout the trial. Patients also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline.
- Arm II (Gemcitabine Hydrochloride, Erlotinib Hydrochloride): [Closed to accrual 2-28-2014.] Patients receive gemcitabine hydrochloride IV over 30 minutes once a week for 3 weeks then off 1 week and erlotinib hydrochloride PO once daily on days 1-28. Treatment repeats every 28 days for up to 5 courses in the absence of disease progression or unacceptable toxicity. Patients undergo CT, MRI, and/or x-ray imaging throughout the trial. Patients also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline.
- Arm III (Chemotherapy): Patients receive the same treatment as in arm I or arm II for one month. Patients undergo CT, MRI, and/or x-ray imaging throughout the trial. Patients also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline.
- Arm IV (Chemotherapy, Chemoradiotherapy): Patients receive the same treatment as in arm I or arm II for one month. Beginning within 7-21 days after completion of chemotherapy, patients undergo radiotherapy (3-dimensional conformal radiotherapy or intensity modulated radiotherapy) 5 days per week for 5.5 weeks (28 fractions). During radiotherapy, patients receive either capecitabine PO twice a day (BID) 5 days per week or fluorouracil IV continuously for 5.5 weeks or until radiotherapy is completed. Patients undergo CT, MRI, and/or x-ray imaging throughout the trial. Patients also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline.
Period: First Step
Arm/Group | Arm I (Gemcitabine Hydrochloride or Combination Chemotherapy) | Arm II (Gemcitabine Hydrochloride, Erlotinib Hydrochloride) | Arm III (Chemotherapy) | Arm IV (Chemotherapy, Chemoradiotherapy)
Started | 379 | 167 | 0 | 0
Randomized to Arm I or Arm II (Closed 02-28-2014.) | 169 | 167 | 0 | 0
Registered to Arm 1 Only (Started 04-02-2014, and as of 06-28-2016, combination chemotherapy was allowed.) | 210 | 0 | 0 | 0
Eligible | 363 | 159 | 0 | 0
Phase II Analysis Population (Randomized to first step and eligible.) | 163 | 159 | 0 | 0
Phase II AE Population (Randomized to first step, eligible, and started protocol treatment.) | 160 | 158 | 0 | 0
Randomized to Arm III | 124 | 50 | 0 | 0
Randomized to Arm IV | 130 | 50 | 0 | 0
Completed (Participants who continued to second step randomization, which requires starting the 5th cycle of the first step treatment and having no progression detected on the 5th cycle CT/MRI.) | 254 | 100 | 0 | 0
Not Completed | 125 | 67 | 0 | 0
Not completed — Withdrawal by Subject | 36 | 19 | 0 | 0
Not completed — Progression | 58 | 23 | 0 | 0
Not completed — Did not start 5th cycle of first step treatment | 15 | 10 | 0 | 0
Not completed — Death | 3 | 4 | 0 | 0
Not completed — Adverse Event | 9 | 5 | 0 | 0
Not completed — Other | 4 | 6 | 0 | 0
Period: Second Step
Arm/Group | Arm I (Gemcitabine Hydrochloride or Combination Chemotherapy) | Arm II (Gemcitabine Hydrochloride, Erlotinib Hydrochloride) | Arm III (Chemotherapy) | Arm IV (Chemotherapy, Chemoradiotherapy)
Started | 0 | 0 | 174 | 180
Phase III Analysis Population (Randomized to second step (Arm III and Arm IV).) | 0 | 0 | 174 | 180
Phase III AE Population (Randomized to second step, and started protocol treatment.) | 0 | 0 | 174 | 180
Completed (Contributed any data to phase III analysis or adverse event reporting.) | 0 | 0 | 174 | 180
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Arm 1 and Arm 2: Phase II analysis population = eligible randomized Step 1 participants.
  Arm 3 and Arm 4: Phase III analysis population = randomized Step 2 participants.
  Phase II and phase III components are reported separately for clarity and so that totals can be seen for each component. Note that 354 participants were in both components.
Groups:
- Arm IV (Chemotherapy, Chemoradiotherapy): Patients receive the same treatment as in arm I or arm II for one month. Beginning within 7-21 days after completion of chemotherapy, patients undergo radiotherapy (3-dimensional conformal radiotherapy or intensity-modulated radiotherapy) 5 days per week for 5.5 weeks (28 fractions). During radiotherapy, patients receive either capecitabine PO BID 5 days per week or fluorouracil IV continuously for 5.5 weeks or until radiotherapy is completed. Patients undergo CT, MRI, and/or x-ray imaging throughout the trial. Patients also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline.
- Total: Total of all reporting groups
Arm/Group | Arm I (Gemcitabine Hydrochloride or Combination Chemotherapy) | Arm II (Gemcitabine Hydrochloride, Erlotinib Hydrochloride) | Arm III (Chemotherapy) | Arm IV (Chemotherapy, Chemoradiotherapy) | Total
Number analyzed (Participants) | 163 | 159 | 174 | 180 | 676
Age, Customized [Count of Participants; unit: Participants] — Population: Baseline characteristics are reported separately for phase II and phase III components.
  Participants
    Phase II Analysis: number analyzed (Participants) | 163 | 159 | 0 | 0 | 322
    Phase II Analysis: ≤ 49 | 18 | 17 |  |  | 35
    Phase II Analysis: 50 - 59 | 42 | 37 |  |  | 79
    Phase II Analysis: 60 - 69 | 57 | 59 |  |  | 116
    Phase II Analysis: 70 - 79 | 35 | 41 |  |  | 76
    Phase II Analysis: ≥ 80 | 11 | 5 |  |  | 16
    Phase III analysis: number analyzed (Participants) | 0 | 0 | 174 | 180 | 354
    Phase III analysis: ≤ 49 |  |  | 17 | 16 | 33
    Phase III analysis: 50 - 59 |  |  | 44 | 44 | 88
    Phase III analysis: 60 - 69 |  |  | 63 | 72 | 135
    Phase III analysis: 70 - 79 |  |  | 43 | 40 | 83
    Phase III analysis: ≥ 80 |  |  | 7 | 8 | 15
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics are reported separately for phase II and phase III components.
  Participants
    Phase II analysis: number analyzed (Participants) | 163 | 159 | 0 | 0 | 322
    Phase II analysis: Female | 75 | 63 |  |  | 138
    Phase II analysis: Male | 88 | 96 |  |  | 184
    Phase III analysis: number analyzed (Participants) | 0 | 0 | 174 | 180 | 354
    Phase III analysis: Female |  |  | 74 | 85 | 159
    Phase III analysis: Male |  |  | 100 | 95 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics are reported separately for phase II and phase III components.
  Participants
    Phase II analysis: number analyzed (Participants) | 163 | 159 | 0 | 0 | 322
    Phase II analysis: Hispanic or Latino | 10 | 8 |  |  | 18
    Phase II analysis: Not Hispanic or Latino | 143 | 143 |  |  | 286
    Phase II analysis: Unknown or Not Reported | 10 | 8 |  |  | 18
    Phase III analysis: number analyzed (Participants) | 0 | 0 | 174 | 180 | 354
    Phase III analysis: Hispanic or Latino |  |  | 10 | 14 | 24
    Phase III analysis: Not Hispanic or Latino |  |  | 158 | 162 | 320
    Phase III analysis: Unknown or Not Reported |  |  | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics are reported separately for phase II and phase III components.
  Participants
    Phase II analysis: number analyzed (Participants) | 163 | 159 | 0 | 0 | 322
    Phase II analysis: American Indian or Alaska Native | 0 | 1 |  |  | 1
    Phase II analysis: Asian | 4 | 4 |  |  | 8
    Phase II analysis: Native Hawaiian or Other Pacific Islander | 1 | 0 |  |  | 1
    Phase II analysis: Black or African American | 10 | 22 |  |  | 32
    Phase II analysis: White | 144 | 129 |  |  | 273
    Phase II analysis: More than one race | 0 | 0 |  |  | 0
    Phase II analysis: Unknown or Not Reported | 4 | 3 |  |  | 7
    Phase III analysis: number analyzed (Participants) | 0 | 0 | 174 | 180 | 354
    Phase III analysis: American Indian or Alaska Native |  |  | 1 | 1 | 2
    Phase III analysis: Asian |  |  | 4 | 8 | 12
    Phase III analysis: Native Hawaiian or Other Pacific Islander |  |  | 0 | 2 | 2
    Phase III analysis: Black or African American |  |  | 19 | 27 | 46
    Phase III analysis: White |  |  | 147 | 139 | 286
    Phase III analysis: More than one race |  |  | 0 | 0 | 0
    Phase III analysis: Unknown or Not Reported |  |  | 3 | 3 | 6
Tumor size largest dimension [Median (Full Range); unit: centimeters] — From pathologic specimen. Population: Baseline characteristics are reported separately for phase II and phase III components.
  centimeters
    Phase II analysis: number analyzed (Participants) | 163 | 159 | 0 | 0 | 322
    Phase II analysis | 3.0 [1.0 to 7.5] | 3.0 [1.0 to 7.6] |  |  | 3.0 [1.0 to 7.6]
    Phase III analysis: number analyzed (Participants) | 0 | 0 | 174 | 180 | 354
    Phase III analysis |  |  | 3.0 [0.9 to 7.9] | 3.0 [1.0 to 6.5] | 3.0 [0.9 to 7.9]
Zubrod Performance Status [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound; 5 = Death Population: Baseline characteristics are reported separately for phase II and phase III components.
  Participants
    Phase II analysis: number analyzed (Participants) | 163 | 159 | 0 | 0 | 322
    Phase II analysis: 0 | 65 | 78 |  |  | 143
    Phase II analysis: 1 | 98 | 81 |  |  | 179
    Phase III analysis: number analyzed (Participants) | 0 | 0 | 174 | 180 | 354
    Phase III analysis: 0 |  |  | 72 | 83 | 155
    Phase III analysis: 1 |  |  | 102 | 97 | 199
Histologic Type [Count of Participants; unit: Participants] — A description of a tumor based on how the cancer cells and tissue look under a microscope. Population: Baseline characteristics are reported separately for phase II and phase III components.
  Participants
    Phase II analysis: number analyzed (Participants) | 163 | 159 | 0 | 0 | 322
    Phase II analysis: Adenocarcinoma | 154 | 153 |  |  | 307
    Phase II analysis: Intraductal papillary mucinous neoplasm with invasive adenocarcinoma | 9 | 6 |  |  | 15
    Phase III analysis: number analyzed (Participants) | 0 | 0 | 174 | 180 | 354
    Phase III analysis: Adenocarcinoma |  |  | 166 | 172 | 338
    Phase III analysis: Intraductal papillary mucinous neoplasm with invasive adenocarcinoma |  |  | 8 | 8 | 16
Pathologic T-Stage [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 6th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. Population: Baseline characteristics are reported separately for phase II and phase III components.
  Participants
    Phase II analysis: number analyzed (Participants) | 163 | 159 | 0 | 0 | 322
    Phase II analysis: T1 | 7 | 8 |  |  | 15
    Phase II analysis: T2 | 30 | 25 |  |  | 55
    Phase II analysis: T3 | 126 | 126 |  |  | 252
    Phase III analysis: number analyzed (Participants) | 0 | 0 | 174 | 180 | 354
    Phase III analysis: T1 |  |  | 2 | 12 | 14
    Phase III analysis: T2 |  |  | 27 | 25 | 52
    Phase III analysis: T3 |  |  | 145 | 143 | 288
Pathologic N-Stage [Count of Participants; unit: Participants] — Regional lymph nodes staging per American Joint Committee on Cancer (AJCC) 6th ed. refers to the number and/or extent of spread of lymph nodes that contain cancer. N0 means lymph nodes aren't involved. A higher number means the cancer is in more lymph nodes, farther away from the original tumor. Population: Baseline characteristics are reported separately for phase II and phase III components.
  Participants
    Phase II analysis: number analyzed (Participants) | 163 | 159 | 0 | 0 | 322
    Phase II analysis: N0 | 45 | 40 |  |  | 85
    Phase II analysis: N1 | 118 | 119 |  |  | 237
    Phase III analysis: number analyzed (Participants) | 0 | 0 | 174 | 180 | 354
    Phase III analysis: N0 |  |  | 42 | 49 | 91
    Phase III analysis: N1 |  |  | 132 | 131 | 263
Number of Positive Lymph Nodes [Count of Participants; unit: Participants] — Population: Baseline characteristics are reported separately for phase II analysis and phase III analysis.
  Participants
    Phase II analysis: number analyzed (Participants) | 163 | 159 | 0 | 0 | 322
    Phase II analysis: 0 | 45 | 40 |  |  | 85
    Phase II analysis: 1-3 | 76 | 78 |  |  | 154
    Phase II analysis: >3 | 42 | 41 |  |  | 83
    Phase III analysis: number analyzed (Participants) | 0 | 0 | 174 | 180 | 354
    Phase III analysis: 0 |  |  | 42 | 49 | 91
    Phase III analysis: 1-3 |  |  | 95 | 79 | 174
    Phase III analysis: >3 |  |  | 37 | 52 | 89
Carbohydrate antigen 19-9 (CA19-9) Level [Count of Participants; unit: Participants] — CA 19-9 is a protein found on the surface of some cancer cells, and is also known as sialyl-Lewis A. It is a tumor marker that is commonly used to help diagnose, manage, and predict pancreatic ductal adenocarcinoma (PDAC). CA 19-9 levels are determined by a blood test and are often elevated in patients with advanced pancreatic cancer. Population: Baseline characteristics are reported separately for phase II and phase III components.
  Participants
    Phase II analysis: number analyzed (Participants) | 163 | 159 | 0 | 0 | 322
    Phase II analysis: ≤ 90 | 152 | 148 |  |  | 300
    Phase II analysis: >90-180 | 11 | 11 |  |  | 22
    Phase III analysis: number analyzed (Participants) | 0 | 0 | 174 | 180 | 354
    Phase III analysis: ≤ 90 |  |  | 163 | 177 | 340
    Phase III analysis: >90-180 |  |  | 11 | 3 | 14
Surgical margins [Count of Participants; unit: Participants] — Population: Baseline characteristics are reported separately for phase II and phase III components.
  Participants
    Phase II analysis: number analyzed (Participants) | 163 | 159 | 0 | 0 | 322
    Phase II analysis: Positive | 27 | 26 |  |  | 53
    Phase II analysis: Negative | 136 | 133 |  |  | 269
    Phase III analysis: number analyzed (Participants) | 0 | 0 | 174 | 180 | 354
    Phase III analysis: Positive |  |  | 30 | 29 | 59
    Phase III analysis: Negative |  |  | 144 | 151 | 295
Type of surgery (phase III only) [Count of Participants; unit: Participants] — Population: Baseline characteristics are reported separately for phase II and phase III components.
  Participants
    Phase II analysis: number analyzed (Participants) | 163 | 159 | 0 | 0 | 322
    Phase II analysis: Classic Pancreaticoduodenectomy (Whipple) | 123 | 117 |  |  | 240
    Phase II analysis: Pylorus preserving pancreaticoduodenectomy | 40 | 40 |  |  | 80
    Phase II analysis: Other | 0 | 2 |  |  | 2
    Phase III analysis: number analyzed (Participants) | 0 | 0 | 174 | 180 | 354
    Phase III analysis: Classic Pancreaticoduodenectomy (Whipple) |  |  | 121 | 139 | 260
    Phase III analysis: Pylorus preserving pancreaticoduodenectomy |  |  | 52 | 41 | 93
    Phase III analysis: Other |  |  | 1 | 0 | 1
Adjuvant Systemic Treatment (Phase III only) [Count of Participants; unit: Participants] — Population: Not reported for phase II analysis.
  Participants
    number analyzed (Participants) | 0 | 0 | 174 | 180 | 354
    Gemcitabine alone |  |  | 116 | 120 | 236
    Gemcitabine + Erlotinib |  |  | 50 | 50 | 100
    Non-oxaliplatin gemcitabine combinations |  |  | 8 | 10 | 18
    FOLFIRINOX or mFOLFIRINOX |  |  | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (Percentage of Participants Alive) [Phase II]
Description: Overall survival is estimated by the Kaplan-Meier method. Survival time is measured from step 1 randomization to date of death from any cause or last known follow-up (censored). Analysis was to occur after 200 deaths were reported.
Time Frame: From step 1 randomization (gemcitabine vs. gemcitabine/erlotinib) to death or last follow-up. Maximum follow-up at the time of the phase II analysis was 6.2 years.
Population: Eligible participants randomized at step 1.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm I (Gemcitabine Hydrochloride or Combination Chemotherapy): Patients receive either gemcitabine hydrochloride or [starting 6-28-2016] allowable combination chemotherapy per standard of care for 5 months. Patients undergo CT, MRI, and/or x-ray imaging throughout the trial. Patients also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline.
- Arm II (Gemcitabine Hydrochloride, Erlotinib Hydrochloride): [Closed to accrual 2-28-14.] Patients receive gemcitabine hydrochloride IV over 30 minutes once a week for 3 weeks then off 1 week and erlotinib hydrochloride PO once daily on days 1-28. Treatment repeats every 28 days for up to 5 courses in the absence of disease progression or unacceptable toxicity. Patients undergo CT, MRI, and/or x-ray imaging throughout the trial. Patients also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline.
Arm/Group | Arm I (Gemcitabine Hydrochloride or Combination Chemotherapy) | Arm II (Gemcitabine Hydrochloride, Erlotinib Hydrochloride)
Number analyzed (Participants) | 163 | 159
months | 29.9 [21.7 to 33.4] | 28.1 [20.7 to 30.9]
Statistical Analysis 1: Comparison: Arm I (Gemcitabine Hydrochloride or Combination Chemotherapy) vs Arm II (Gemcitabine Hydrochloride, Erlotinib Hydrochloride); A total of 200 deaths between the arms will provide 80% power to detect a signal for an increase in median overall survival from 22 to 28.8 months and 90% power to detect a signal for an increase in median overall survival from 22 to 30.6 months (HRs of 0.76 and 0.72, respectively, in favor of the erlotinib arm) with the addition of erlotinib and a 1-sided alpha of 0.15; Test type: Superiority; p = 0.62, Log Rank — One-sided significance level = 0.15; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.79 to 1.38] — Reference level = Arm I

2. Primary Outcome: Overall Survival (Percentage of Participants Alive) [Phase III]
Description: Overall survival (OS) is estimated by the Kaplan-Meier method. Survival time is measured from step 2 randomization to date of death from any cause or last known follow-up (censored). Analysis was to occur at the earlier of 316 reported deaths or when all patients have five years potential follow-up from step 2 randomization.
Time Frame: From step 2 randomization (chemotherapy vs. chemotherapy followed by chemoradiation) to the date of death or last follow-up. Maximum follow-up at time of the phase III analysis was 12.8 years, measured from step 2 randomization.
Population: Participants randomized at step 2.
Measure: Median (90% Confidence Interval); unit: months
Groups:
- Arm IV (Chemotherapy, Chemoradiotherapy): Patients receive the same treatment as in arm I or arm II for one month. Beginning within 7-21 days after completion of chemotherapy, patients undergo radiotherapy (RT) (3-dimensional conformal radiotherapy or intensity modulated radiotherapy) 5 days per week for 5.5 weeks (28 fractions). During radiotherapy, patients receive either capecitabine PO BID 5 days per week or fluorouracil IV continuously for 5.5 weeks or until radiotherapy is completed. Patients undergo CT, MRI, and/or x-ray imaging throughout the trial. Patients also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline.
Arm/Group | Arm III (Chemotherapy) | Arm IV (Chemotherapy, Chemoradiotherapy)
Number analyzed (Participants) | 174 | 180
months | 31.1 [25.3 to 37.6] | 27.3 [24.5 to 31.7]
Statistical Analysis 1: Comparison: Arm III (Chemotherapy) vs Arm IV (Chemotherapy, Chemoradiotherapy); 316 deaths from step 2 randomized patients provides 80% power, with 0.05 1-sided alpha, to detect an OS increase (HR=0.76 in favor of arm IV), corresponding to increasing median OS from 17 to 22.5 months with the addition of RT. For analysis triggered by patients having 5 years potential follow-up from step 2 randomization, it is projected that at least 265 events will be observed, providing at least 72% power. The trigger used for the primary analysis was 5-years of follow-up (270 deaths); Test type: Superiority; p = 0.38, Log Rank — One-sided significance level = 0.05; Hazard Ratio (HR) = 0.96, 90% CI 2-sided [0.79 to 1.18] — Reference level = Arm III

3. Secondary Outcome: Disease-free Survival (Percentage of Participants Alive Without Disease) [Phase II]
Description: Disease-free survival is estimated by the Kaplan-Meier method. Disease-free survival time is measured from step 1 randomization to the first date of local or regional disease, distant metastases, second primary tumor, death due to any cause, or last known follow-up (censored). Analysis was to occur after 200 deaths were reported.
Time Frame: From step1 randomization (gemcitabine vs. gemcitabine/erlotinib) to disease event, death, or last follow-up. Maximum follow-up at the time of the phase II analysis was 6.2 years.
Population: Eligible participants randomized at step 1.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Gemcitabine Hydrochloride or Combination Chemotherapy) | Arm II (Gemcitabine Hydrochloride, Erlotinib Hydrochloride)
Number analyzed (Participants) | 163 | 159
months | 12.7 [10.8 to 15.7] | 12.4 [9.7 to 16.5]
Statistical Analysis 1: Comparison: Arm I (Gemcitabine Hydrochloride or Combination Chemotherapy) vs Arm II (Gemcitabine Hydrochloride, Erlotinib Hydrochloride); Test type: Superiority; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.80 to 1.31] — Reference level = Arm I

4. Secondary Outcome: Disease-free Survival (Percentage of Participants Alive Without Disease) [Phase III]
Description: Disease-free survival is estimated by the Kaplan-Meier method. Disease-free survival time is measured from step 2 randomization to the first date of local or regional disease, distant metastases, second primary tumor, death due to any cause, or last known follow-up (censored). Analysis was to occur at the earlier of 316 reported deaths or when all participants have five years potential follow-up from second step randomization.
Time Frame: From step 2 randomization (chemotherapy vs. chemotherapy followed by chemoradiation) to disease event, death, or last follow-up. Maximum follow-up at time of the phase III analysis was 12.8 years, measured from step 2 randomization.
Population: Participants randomized at step 2.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm III (Chemotherapy) | Arm IV (Chemotherapy, Chemoradiotherapy)
Number analyzed (Participants) | 174 | 180
months | 12.4 [9.6 to 15.2] | 15.6 [13.2 to 18.8]
Statistical Analysis 1: Comparison: Arm III (Chemotherapy) vs Arm IV (Chemotherapy, Chemoradiotherapy); Test type: Superiority; Hazard Ratio (HR) = 0.82, 90% CI 2-sided [0.68 to 0.99] — Reference level = Arm III

5. Secondary Outcome: Number of Participants by Highest Grade Adverse Event Reported (Phase II)
Description: Assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 which grades adverse event severity from 1=mild to 5=death. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: as for outcome 1
Population: Eligible participants randomized in Step 1 who started protocol treatment and were assessed for adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Gemcitabine Hydrochloride or Combination Chemotherapy) | Arm II (Gemcitabine Hydrochloride, Erlotinib Hydrochloride)
Number analyzed (Participants) | 160 | 158
Participants
  Grade 1 | 6 | 3
  Grade 2 | 20 | 24
  Grade 3 | 100 | 101
  Grade 4 | 32 | 27
  Grade 5 | 2 | 3

6. Secondary Outcome: Number of Participants by Highest Grade Adverse Event Reported (Phase III)
Description: Assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 which grades adverse event severity from 1=mild to 5=death.
Time Frame: From step 2 randomization (chemotherapy vs. chemotherapy followed by chemoradiation) to death or last follow-up. Maximum follow-up at time of the phase III analysis was 12.8 years, measured from step 2 randomization.
Population: Participants randomized at step 2.
Measure: Count of Participants; unit: Participants
Groups:
- Arm IV (Chemotherapy, Chemoradiotherapy): Patients receive the same treatment as in arm I or arm II for one month. Beginning within 7-21 days after completion of chemotherapy, patients undergo radiotherapy (3-dimensional conformal radiotherapy or intensity modulated radiotherapy) 5 days per week for 5.5 weeks (28 fractions). During radiotherapy, patients receive either capecitabine PO BID 5 days per week or fluorouracil IV continuously for 5.5 weeks or until radiotherapy is completed. Patients undergo CT, MRI, and/or x-ray imaging throughout the trial. Patients also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline.
Arm/Group | Arm III (Chemotherapy) | Arm IV (Chemotherapy, Chemoradiotherapy)
Number analyzed (Participants) | 174 | 180
Participants
  Grade 1 | 22 | 16
  Grade 2 | 50 | 56
  Grade 3 | 67 | 79
  Grade 4 | 21 | 23
  Grade 5 | 1 | 1

7. Secondary Outcome: Frequency of Objective Criteria of Resectability as Measured by Preoperative Imaging
Time Frame: Baseline
Reporting Status: Not Posted, anticipated posting 2025-12

8. Secondary Outcome: Overall Survival by Baseline Fatigue Group
Description: Overall survival is estimated by the Kaplan-Meier method. Survival time is measured from step 1 randomization to date of death from any cause or last known follow-up (censored). Baseline fatigue is measured by Functional Assessment of Chronic Illness Therapy-Fatigue (FACT-F) questionnaire which has a range of 0 to 52 with a higher score indicating less fatigue. Patients with low fatigue at baseline (FACIT-F score > 30) will be compared to patients with high fatigue at baseline (FACIT-F scores ≤ 30). The analysis population is all enrolled eligible participants who consented to the quality of life study component and who have baseline FACT-F data.
Time Frame: From enrollment to death or last follow-up.
Reporting Status: Not Posted, anticipated posting 2025-12

9. Other Pre Specified Outcome: Determination of National Institutes of Health (NIH) Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue and Overall Survival
Description: Baseline PROMIS Fatigue scores will be analyzed to determine if there is a cut point (adjusting for multiple comparisons) that correlates with overall survival using the log-rank statistic. The analysis population is all enrolled eligible participants who consented to the quality of life study component and who have baseline PROMIS data.
Time Frame: From enrollment to death or last follow-up.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Arms I and II: From step 1 randomization (gemcitabine versus vs. gemcitabine/erlotinib) to the date of last follow-up. Maximum follow-up at the time of the phase II analysis was 6.2 years. Arms III and IV: From the date of enrollment to the date of last follow-up. Maximum follow-up at time of phase III analysis was 13.2 years.
Description: Note that adverse events from Arm I and II participants who continued to step 2 randomization will also appear in the adverse events for Arms III and IV.
Groups:
- Arm I (Gemcitabine Hydrochloride or Combination Chemotherapy): Participants receive either gemcitabine hydrochloride or [starting 06-28-2016] allowable combination chemotherapy per standard of care for 5 months. Participants undergo CT, MRI, and/or x-ray imaging throughout the trial. Participants also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline.
- Arm II (Gemcitabine Hydrochloride, Erlotinib Hydrochloride): [Closed to accrual 2-28-2014.] Participants receive gemcitabine hydrochloride IV over 30 minutes once a week for 3 weeks then off 1 week and erlotinib hydrochloride PO once daily on days 1-28. Treatment repeats every 28 days for up to 5 courses in the absence of disease progression or unacceptable toxicity. Participants undergo CT, MRI, and/or x-ray imaging throughout the trial. Participants also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline.
- Arm III (Chemotherapy): Participants receive the same treatment as in arm I or arm II for one month. Participants undergo CT, MRI, and/or x-ray imaging throughout the trial. Participants also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline.
- Arm IV (Chemotherapy, Chemoradiotherapy): Participants receive the same treatment as in arm I or arm II for one month. Beginning within 7-21 days after completion of chemotherapy, Participants undergo radiotherapy (3-dimensional conformal radiotherapy or intensity-modulated radiotherapy) 5 days per week for 5.5 weeks (28 fractions). During radiotherapy, Participants receive either capecitabine PO BID 5 days per week or fluorouracil IV continuously for 5.5 weeks or until radiotherapy is completed. Participants undergo CT, MRI, and/or x-ray imaging throughout the trial. Participants also undergo blood sample collection during screening and follow-up and undergo tissue sample collection at baseline.
Arm/Group | Arm I (Gemcitabine Hydrochloride or Combination Chemotherapy) | Arm II (Gemcitabine Hydrochloride, Erlotinib Hydrochloride) | Arm III (Chemotherapy) | Arm IV (Chemotherapy, Chemoradiotherapy)
All-Cause Mortality (participants affected / at risk) | 103/160 | 100/158 | 136/174 | 134/180
Serious Adverse Events (participants affected / at risk) | 38/160 | 45/158 | 33/174 | 31/180
Other Adverse Events (participants affected / at risk) | 158/160 | 157/158 | 173/174 | 179/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Gemcitabine Hydrochloride or Combination Chemotherapy) (N=160) | Arm II (Gemcitabine Hydrochloride, Erlotinib Hydrochloride) (N=158) | Arm III (Chemotherapy) (N=174) | Arm IV (Chemotherapy, Chemoradiotherapy) (N=180)
Anemia (Blood and lymphatic system disorders) | 3 | 9 | 5 | 3
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 1 | 1 | 2
Heart failure (Cardiac disorders) | 1 | 1 | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2 | 1 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 6 | 7 | 5
Ascites (Gastrointestinal disorders) | 1 | 1 | 2 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 4 | 1 | 4
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Jejunal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Small intestine ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2 | 1
Chills (General disorders) | 0 | 1 | 1 | 0
Death NOS (General disorders) | 0 | 1 | 0 | 0
Edema limbs (General disorders) | 3 | 1 | 0 | 1
Fatigue (General disorders) | 2 | 5 | 4 | 2
Fever (General disorders) | 1 | 7 | 4 | 3
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 2 | 1 | 0
Irritability (General disorders) | 0 | 1 | 0 | 1
Localized edema (General disorders) | 1 | 0 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1 | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 1 | 1 | 0
Biliary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Bladder infection (Infections and infestations) | 1 | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Hepatic infection (Infections and infestations) | 0 | 1 | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 3 | 4 | 2 | 1
Infective myositis (Infections and infestations) | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 3 | 3 | 3 | 3
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 3 | 5 | 1 | 4
Skin infection (Infections and infestations) | 2 | 2 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 4 | 4 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 1
Small intestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 0
Cardiac troponin I increased (Investigations) | 0 | 1 | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 1 | 0 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1 | 1 | 0
INR increased (Investigations) | 0 | 2 | 0 | 0
Investigations - Other, specify (Investigations) | 0 | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 4 | 6 | 4 | 1
Platelet count decreased (Investigations) | 1 | 2 | 3 | 0
Weight loss (Investigations) | 0 | 3 | 2 | 1
White blood cell decreased (Investigations) | 2 | 1 | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 3 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 5 | 2 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 4 | 2 | 2 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 1
Stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 3 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 2 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 2
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 2 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 1 | 3 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 3 | 2 | 3 | 0
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Gemcitabine Hydrochloride or Combination Chemotherapy) (N=160) | Arm II (Gemcitabine Hydrochloride, Erlotinib Hydrochloride) (N=158) | Arm III (Chemotherapy) (N=174) | Arm IV (Chemotherapy, Chemoradiotherapy) (N=180)
Anemia (Blood and lymphatic system disorders) | 122 | 119 | 139 | 142
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 10 | 11 | 11 | 11
Blurred vision (Eye disorders) | 6 | 5 | 12 | 7
Abdominal distension (Gastrointestinal disorders) | 11 | 7 | 8 | 6
Abdominal pain (Gastrointestinal disorders) | 66 | 69 | 74 | 85
Ascites (Gastrointestinal disorders) | 14 | 10 | 9 | 13
Bloating (Gastrointestinal disorders) | 13 | 18 | 13 | 22
Constipation (Gastrointestinal disorders) | 42 | 40 | 64 | 48
Diarrhea (Gastrointestinal disorders) | 89 | 90 | 87 | 112
Dry mouth (Gastrointestinal disorders) | 7 | 15 | 20 | 8
Dyspepsia (Gastrointestinal disorders) | 23 | 32 | 29 | 24
Flatulence (Gastrointestinal disorders) | 9 | 13 | 13 | 25
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 | 6 | 9 | 11
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 16 | 11 | 13 | 19
Mucositis oral (Gastrointestinal disorders) | 22 | 24 | 20 | 24
Nausea (Gastrointestinal disorders) | 109 | 90 | 111 | 119
Vomiting (Gastrointestinal disorders) | 45 | 48 | 47 | 48
Chills (General disorders) | 16 | 22 | 28 | 20
Edema limbs (General disorders) | 46 | 41 | 47 | 59
Fatigue (General disorders) | 123 | 121 | 135 | 147
Fever (General disorders) | 43 | 33 | 48 | 46
Flu like symptoms (General disorders) | 8 | 9 | 13 | 12
Localized edema (General disorders) | 8 | 4 | 6 | 10
Pain (General disorders) | 39 | 29 | 39 | 46
Sepsis (Infections and infestations) | 7 | 5 | 9 | 7
Skin infection (Infections and infestations) | 3 | 9 | 9 | 11
Upper respiratory infection (Infections and infestations) | 8 | 2 | 5 | 6
Urinary tract infection (Infections and infestations) | 11 | 14 | 13 | 11
Alanine aminotransferase increased (Investigations) | 58 | 57 | 57 | 67
Alkaline phosphatase increased (Investigations) | 56 | 53 | 53 | 64
Aspartate aminotransferase increased (Investigations) | 64 | 73 | 68 | 73
Blood bilirubin increased (Investigations) | 18 | 20 | 16 | 15
Creatinine increased (Investigations) | 15 | 18 | 19 | 16
Investigations - Other, specify (Investigations) | 5 | 7 | 9 | 12
Lymphocyte count decreased (Investigations) | 34 | 27 | 29 | 47
Neutrophil count decreased (Investigations) | 99 | 82 | 99 | 113
Platelet count decreased (Investigations) | 96 | 75 | 87 | 108
Weight gain (Investigations) | 6 | 8 | 16 | 5
Weight loss (Investigations) | 40 | 34 | 44 | 44
White blood cell decreased (Investigations) | 74 | 78 | 76 | 88
Anorexia (Metabolism and nutrition disorders) | 61 | 61 | 66 | 66
Dehydration (Metabolism and nutrition disorders) | 19 | 14 | 13 | 17
Hyperglycemia (Metabolism and nutrition disorders) | 63 | 59 | 60 | 69
Hyperkalemia (Metabolism and nutrition disorders) | 10 | 10 | 10 | 15
Hypernatremia (Metabolism and nutrition disorders) | 9 | 14 | 9 | 16
Hypoalbuminemia (Metabolism and nutrition disorders) | 61 | 54 | 59 | 58
Hypocalcemia (Metabolism and nutrition disorders) | 42 | 39 | 36 | 39
Hypoglycemia (Metabolism and nutrition disorders) | 9 | 13 | 11 | 8
Hypokalemia (Metabolism and nutrition disorders) | 34 | 41 | 43 | 39
Hypomagnesemia (Metabolism and nutrition disorders) | 10 | 10 | 14 | 9
Hyponatremia (Metabolism and nutrition disorders) | 26 | 29 | 28 | 32
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3 | 9 | 8 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 5 | 16 | 16
Arthritis (Musculoskeletal and connective tissue disorders) | 5 | 5 | 10 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 34 | 23 | 34 | 29
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 6 | 9
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 16 | 20 | 25 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 8 | 21 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 10 | 18 | 18
Dizziness (Nervous system disorders) | 20 | 25 | 31 | 28
Dysgeusia (Nervous system disorders) | 17 | 22 | 33 | 20
Headache (Nervous system disorders) | 23 | 28 | 33 | 41
Paresthesia (Nervous system disorders) | 8 | 7 | 8 | 12
Peripheral motor neuropathy (Nervous system disorders) | 2 | 8 | 6 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 19 | 25 | 32 | 31
Anxiety (Psychiatric disorders) | 19 | 15 | 22 | 17
Depression (Psychiatric disorders) | 17 | 15 | 18 | 13
Insomnia (Psychiatric disorders) | 27 | 23 | 37 | 28
Proteinuria (Renal and urinary disorders) | 3 | 5 | 9 | 2
Urinary frequency (Renal and urinary disorders) | 4 | 8 | 14 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 16 | 30 | 30
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 34 | 32 | 35 | 39
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 | 7 | 5 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 18 | 27 | 38 | 24
Dry skin (Skin and subcutaneous tissue disorders) | 13 | 30 | 29 | 18
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 10 | 10 | 24
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 20 | 26 | 12
Rash acneiform (Skin and subcutaneous tissue disorders) | 7 | 74 | 36 | 33
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 | 42 | 28 | 27
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 16 | 17 | 12 | 16
Hypertension (Vascular disorders) | 11 | 16 | 20 | 25
Hypotension (Vascular disorders) | 11 | 7 | 12 | 5
Thromboembolic event (Vascular disorders) | 12 | 17 | 14 | 13

LIMITATIONS AND CAVEATS:
Based on negative results from trial NCT00634725 regarding the question of gemcitabine versus gemcitabine plus erlotinib in locally unresectable pancreatic cancer patients, this study was amended to stop the erlotinib randomization and to change the erlotinib question to a randomized phase II design using the patients already randomized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT01013649/Prot_SAP_000.pdf